CLINICAL TRIAL: NCT01698632
Title: A Multicentre Study to Examine the Short and Long Term Outcomes of the Conservative Management of Benign-looking Adnexal Masses and the Pre-operative Characterisation of Ovarian Tumours
Brief Title: International Ovarian Tumour Analysis (IOTA) Phase 5
Acronym: IOTA-5
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Dirk Timmerman, Prof. Dr. Dirk Timmerman, KU Leuven
Other Study IDs: IOTA5 S51375/B32220095331; USF IRB Pro00009001 (Other: University of South Florida)
Record Dates: First submitted 2012-09-19; First posted 2012-10-03 (Estimated); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Adnexal Masses; Ovarian Cysts; Ovarian Tumors
Keywords: Adnexal masses; Ovarian cysts; Ovarian tumors
MeSH Terms: conditions — Ovarian Cysts; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- benign-looking adnexal masses

SUMMARY:
The purpose of this study is to learn more about the appearance and behavior of benign-looking adnexal masses.

* Benign-looking means that when viewed here by ultrasound it has the appearance of looking not harmful or not malignant.
* Adnexal refers to the 'adnexa', the space in the female pelvis on either side of the uterus (or where the uterus used to be if you previously had a hysterectomy). The adnexa includes, but is not limited to, the ovaries and the fallopian tubes.
* Masses refers to a variety of structures, including but not limited to:

  * ovarian cysts that are fluid filled sacs within or attached to an ovary
  * ovarian tumors that can be solid tissue or a combination of cysts and solid tissue
  * hydrosalpinges that are fluid collections in the fallopian tube

Many women have what appear to be benign adnexal masses. Many times, removal of the masses with surgery is not necessary. Often surgery is performed unnecessarily, for fear that these masses could be cancer. There is not much information available for doctors to know how and when to follow these masses, or which ones will become cancer.

This study will combine information from centers all around the world regarding the behavior of all types of benign adnexal masses. The aim of this study is to develop decision tools for doctors to know the best way to treat these masses in order to improve the detection of ovarian cancer while at the same time reduce the number of unnecessary operations.

ELIGIBILITY:
Inclusion Criteria:

* Any woman at least 18 years old with an adnexal mass.
* Any mass with benign ultrasound morphology may be suitable for conservative management.
* Pregnant patients can be included, but their data will be analysed separately.

Exclusion Criteria:

* Cysts that are deemed to be clearly physiological and less than 3 cm in maximum diameter are not eligible for inclusion.
* Any cyst with features of malignancy is excluded from the conservative management
* The denial or withdrawal of oral informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women being seen for adnexal masses.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Actual)
Dates: Start 2012-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of complications such as rupture, torsion, or malignancy in patients with benign looking conservatively treated masses | Up to five years

SECONDARY OUTCOMES:
Test the published IOTA diagnostic models for predicting that a mass is malignant at first visit or benign | Up to five years
  Also to predict complications (e.g. occurrence of malignancy and other) during long-term follow-up using the diagnostic models

OTHER OUTCOMES:
Investigate factors related to the need for surgery during long-term follow-up | Up to five years
Study natural history of conservatively treated benign-looking adnexal masses | Up to five years
  Also to establish descriptive curves of the longitudinal changes seen in parameters from conservatively managed benign tumors (for example, change in diameter, size of any solid component, number of papillations or color score)

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Timmerman, PhD, Principal Investigator — University Hospitals, KU Leuven
Locations (1):
- USF Health South Tampa Center for Advanced Healthcare, Tampa, Florida, United States

REFERENCES:
- [Derived] Pascual MA, Vancraeynest L, Timmerman S, Ceusters J, Ledger A, Graupera B, Rodriguez I, Valero B, Landolfo C, Testa AC, Bourne T, Timmerman D, Valentin L, Van Calster B, Froyman W. Validation of ADNEX and IOTA two-step strategy and estimation of risk of complications during follow-up of adnexal masses in low-risk population. Ultrasound Obstet Gynecol. 2024 Sep;64(3):395-404. doi: 10.1002/uog.27642. Epub 2024 Aug 16. PMID 38477179
- [Derived] Landolfo C, Ceusters J, Valentin L, Froyman W, Van Gorp T, Heremans R, Baert T, Wouters R, Vankerckhoven A, Van Rompuy AS, Billen J, Moro F, Mascilini F, Neumann A, Van Holsbeke C, Chiappa V, Bourne T, Fischerova D, Testa A, Coosemans A, Timmerman D, Van Calster B. Comparison of the ADNEX and ROMA risk prediction models for the diagnosis of ovarian cancer: a multicentre external validation in patients who underwent surgery. Br J Cancer. 2024 Apr;130(6):934-940. doi: 10.1038/s41416-024-02578-x. Epub 2024 Jan 19. PMID 38243011
- [Derived] Van Calster B, Valentin L, Froyman W, Landolfo C, Ceusters J, Testa AC, Wynants L, Sladkevicius P, Van Holsbeke C, Domali E, Fruscio R, Epstein E, Franchi D, Kudla MJ, Chiappa V, Alcazar JL, Leone FPG, Buonomo F, Coccia ME, Guerriero S, Deo N, Jokubkiene L, Savelli L, Fischerova D, Czekierdowski A, Kaijser J, Coosemans A, Scambia G, Vergote I, Bourne T, Timmerman D. Validation of models to diagnose ovarian cancer in patients managed surgically or conservatively: multicentre cohort study. BMJ. 2020 Jul 30;370:m2614. doi: 10.1136/bmj.m2614. PMID 32732303
- [Derived] Froyman W, Landolfo C, De Cock B, Wynants L, Sladkevicius P, Testa AC, Van Holsbeke C, Domali E, Fruscio R, Epstein E, Dos Santos Bernardo MJ, Franchi D, Kudla MJ, Chiappa V, Alcazar JL, Leone FPG, Buonomo F, Hochberg L, Coccia ME, Guerriero S, Deo N, Jokubkiene L, Kaijser J, Coosemans A, Vergote I, Verbakel JY, Bourne T, Van Calster B, Valentin L, Timmerman D. Risk of complications in patients with conservatively managed ovarian tumours (IOTA5): a 2-year interim analysis of a multicentre, prospective, cohort study. Lancet Oncol. 2019 Mar;20(3):448-458. doi: 10.1016/S1470-2045(18)30837-4. Epub 2019 Feb 5. PMID 30737137

DOCUMENTS (2):
  • Study Protocol (2012-01-23): https://cdn.clinicaltrials.gov/large-docs/32/NCT01698632/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-28): https://cdn.clinicaltrials.gov/large-docs/32/NCT01698632/SAP_002.pdf